CLINICAL TRIAL: NCT02867293
Title: Impact Of Timing Of Drainage Of Massive Ascites On Operative And Post-Operative Course In Living-Donor Liver Transplant Recipients. A Prospective Randomized Controlled Trial.
Acronym: AscitesLDLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, AlRefaey Kandeel, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ascites
Record Dates: First submitted 2016-08-11; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Massive Ascites
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preop-drainage (Active Comparator): ascites drained over the pre-operative week through multiple ultrasound guided paracentesis
  Interventions: Procedure: ultrasound guided ascitic fluid drainage; Device: ultrasound
- Op-drainage (Active Comparator): ascetic fluid drained through an abdominal incision after anesthesia
  Interventions: Procedure: operative drainage of ascites through small skin incision after induction of anesthesia

INTERVENTIONS:
Procedure: ultrasound guided ascitic fluid drainage
  Arms: Preop-drainage
Procedure: operative drainage of ascites through small skin incision after induction of anesthesia
  Arms: Op-drainage
Device: ultrasound
  Arms: Preop-drainage

SUMMARY:
Massive ascites is usually controlled over several weeks pre-operatively in liver transplant recipients with the risk of encephalopathy and peritonitis. We hypothesized that intra-operative drainage of ascites will be safe and avoids the inherent risks of pre-operative drainage.

ELIGIBILITY:
Inclusion Criteria:

* liver transplant candidates with tense acsites

Exclusion Criteria:

* severe coagulpathy (INR more than 2 or platlet count less than 50) MELD more than 20

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
graft survival | one year

SECONDARY OUTCOMES:
patient survival | one year

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Mansoura university, Al Mansurah, Dakahlia Governorate
  - Mansoura university, Al Mansurah, Dkahleya

IPD SHARING:
Plan to Share IPD: Yes